CLINICAL TRIAL: NCT03821298
Title: Psychosocial Factors a Prognostic Study of Pain Persistence in Patients With Thumb Carpometacarpal Osteoarthritis
Brief Title: Psychosocial Factors a Prognostic Study of Pain in Patients With CMC Osteoarthritis
Acronym: CMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gannon University (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Principal Investigator, Kristin Valdes, Assistant Professor of Occupational Therapy, Gannon University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-2018
Record Dates: First submitted 2019-01-26; First posted 2019-01-29 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Pain; Osteoarthritis
Keywords: pain; osteoarthritis; function
MeSH Terms: conditions — Pain; Osteoarthritis | interventions — Orthotic Devices

STUDY DESIGN:
Intervention Model Description: Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of Care (Experimental): short thumb orthoses during ADL, joint reeducation for hand used, radial nerve gliding exercises and thumb proprioception exercises
  Interventions: Other: Standard of Care Hand Therapy

INTERVENTIONS:
Other: Standard of Care Hand Therapy — 8 sessions 2 times a week for 4 weeks
  Other Names: Orthosis; Radial Nerve Gliding; Joint Protection Education; Proprioception exercises

SUMMARY:
In this clinical trial, females with a diagnosis of thumb CMC OA, will be recruited. The primary outcome of potential risk factors of osteoarthritis, pain and function will be measured using the demographic data, visual analog scale (VAS) and Disabilities of the Arm, Shoulder and Hand (QuickDASH). Secondary out-comes will include the Pain Self-Efficacy Questionnaire (PSEQ), Tampa Scale of Kinesiophobia (TSK), Fear Avoidance Beliefs Questionnaire (FABQ), Hospital Anxiety and Depression Scale (HADS) and Impairment and Functioning Inventory (IFI). Measurements will be taken at the baseline, three, six and 12 months follow up.

DETAILED DESCRIPTION:
The study will start recruitment in April 2019.In this clinical trial, 50-100 females, aged 50 to 90 years of age, with a diagnosis of thumb CMC OA, will be recruited. The primary outcome of potential risk factors of osteoarthritis, pain and function will be measured using the demographic data, visual analog scale (VAS) and Disabilities of the Arm, Shoulder and Hand (QuickDASH). Secondary out-comes will include the Pain Self-Efficacy Questionnaire (PSEQ), Tampa Scale of Kinesiophobia (TSK), Fear Avoidance Beliefs Questionnaire (FABQ), Hospital Anxiety and Depression Scale (HADS) and Impairment and Functioning Inventory (IFI). Measurements will be tak-en at the baseline, three, six and 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* women older than 18 years
* diagnosed with bilateral thumb CMC OA
* a reported pain intensity during activities of daily living (ADLs) of up to 4 of 10 on the visual analog scale (VAS)
* The referring hand surgeon will made the diagnosis of CMC OA based on radiographs and clinical exploration.

Exclusion Criteria:

* neurologic disorder affecting the upper limb
* had received previous treatment for their hand problem in the last 6 months including an intra-articular joint injection to wrist, fingers, or thumb
* had fractures or a significant hand injury or previous surgery to the wrist or hand
* had hand or finger tenosynovitis and/or Dupuytren disease
* patients who did not complete any questionnaire or if they did not sign the informed consent.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 12 months Visual Analog Scale (VAS) | baseline, three, six and 12 months follow up
  Pain scale VAS; 0: no pain, 100: maximum pain
Change from baseline to 12 months Quick Disabilities of the Arm, Shoulder and Hand | baseline, three, six and 12 months follow up
  Self Report Function,QuickDash scores range from 0 to 100, higher scores means more dysfunction

SECONDARY OUTCOMES:
Change from baseline to 12 months using the Pain Self-Efficacy Questionnaire | baseline, three, six and 12 months follow up
  Confidence in performing activities of daily living,They answer by circling a number on a 7-point Likert scale under each item, where 0 = not at all confident and 6= completely confident. A total score, ranging from 0 to 60, is calculated by adding the scores for each item. Higher scores reflect stronger self- efficacy beliefs.
Change from baseline to 12 months using the Tampa Scale of Kinesiophobia | baseline, three, six and 12 months follow up
  measure of fear of movement, the total score ranges between 17 and 68. A high value on the TSK indicates a high degree of kinesiophobia, and a cutoff score was developed by Vlaeyen (1995), where a score of 37or over is considered as a high score, while scores below that are considered as low scores. Use of a total score (including all 17 items) is recommended, although practitioners may wish to interpret results using two subscales
Change from baseline to 12 months using the Fear Avoidance Beliefs Questionnaire | baseline, three, six and 12 months follow up
  self report measure of avoidance of activities of daily livin, The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance belief
Change from baseline to 12 months using the Hospital Anxiety and Depression Scale | baseline, three, six and 12 months follow up
  Measure Depression and Anxiety,Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score indicates heightened anxiety or depression
Change in from baseline to 12 months using the Impairment and Functioning Inventory | baseline, three, six and 12 months follow up
  Function, . It consists of 30 items with two related subscales: Daily Functioning and Impairment (perceived current level of functioning compared with the level of functioning before pain onset). 30 questions scored 0-4. Higher score indicates increased ability to perform activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- Gannon University, Ruskin, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pincus T, Burton AK, Vogel S, Field AP. A systematic review of psychological factors as predictors of chronicity/disability in prospective cohorts of low back pain. Spine (Phila Pa 1976). 2002 Mar 1;27(5):E109-20. doi: 10.1097/00007632-200203010-00017. PMID 11880847
- [Result] Kerns RD, Sellinger J, Goodin BR. Psychological treatment of chronic pain. Annu Rev Clin Psychol. 2011;7:411-34. doi: 10.1146/annurev-clinpsy-090310-120430. PMID 21128783
- [Result] Haugen IK, Englund M, Aliabadi P, Niu J, Clancy M, Kvien TK, Felson DT. Prevalence, incidence and progression of hand osteoarthritis in the general population: the Framingham Osteoarthritis Study. Ann Rheum Dis. 2011 Sep;70(9):1581-6. doi: 10.1136/ard.2011.150078. Epub 2011 May 27. PMID 21622766
- [Result] Zhang W, Doherty M, Leeb BF, Alekseeva L, Arden NK, Bijlsma JW, Dincer F, Dziedzic K, Hauselmann HJ, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Maheu E, Martin-Mola E, Pavelka K, Punzi L, Reiter S, Sautner J, Smolen J, Verbruggen G, Zimmermann-Gorska I. EULAR evidence based recommendations for the management of hand osteoarthritis: report of a Task Force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2007 Mar;66(3):377-88. doi: 10.1136/ard.2006.062091. Epub 2006 Oct 17. PMID 17046965